CLINICAL TRIAL: NCT05867628
Title: The Impact of an Intensive Activities-based Locomotor Training Program on Activity Capacity, Performance, and Participation in Children With Cerebral Palsy
Brief Title: Intensive Activities-based Locomotor Training Program in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Other Study IDs: 1922152-2
Record Dates: First submitted 2023-04-17; First posted 2023-05-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; children; activities-based locomotor training; neuroplasticity
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Activities-based locomotor training (physical therapy) — AB-LT is implemented through a combination of partial body weight supported treadmill training, overground walking, and play-based activities.
  Other Names: play-based physical therapy

SUMMARY:
The goal of the proposed work is to investigate the impact of an intensive 3-week activities-based locomotor training (AB-LT) program on activity capacity, activity performance, and participation in children with cerebral palsy (CP). Caregiver perspectives will provide a holistic assessment of the program.

ELIGIBILITY:
Inclusion Criteria:

* Intervention: Participants will be included if they have a diagnosis of CP and are between the ages of 2 to 12 years. They must also be enrolled in the 3-week AB-LT program at Fortis Therapy Center.

Parent Interview: Participants will be included if they are the parent or guardian (any age) of a child who participated in the 3-week AB-LT program and attended at least 3 sessions with their child.

Exclusion Criteria:

* Intervention study: Participants will be excluded if they have had surgery or botulinum toxin injections in the previous 6 months or have uncontrolled epilepsy or cardiovascular disease.

Parent Interview: Participants will be excluded if they have not attended at least 3 AB-LT sessions with their child.

Ages: 2 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-66 (GMFM) | 6.5 months
  Gross Motor Function Measure-66: Items scored on 0-3 scale. Minimum value: 0. Maximum value: 99. Higher scores indicate better outcome.
Pediatric Neuromuscular Recovery Scale (PedsNRS) | 6.5 months
  Pediatric Neuromuscular Recovery Scale: Each of the 13 items on the Peds NRS have 12 phases. Each item is scored on a 12-point scale, with one point allocated to each phase of the item. The age-appropriate item cards instruct the rater to begin at a designated "start phase" indicated by a bold box around the phase within the 12 phases on each card. If the child cannot perform the movement as listed in the start phase (which may be midway through the card), the rater starts at the beginning of the item card and assesses the child's performance at the first phase for that item. The rater continues sequentially through the 12 phases on the card until the child is unable to perform a phase. The rater scores the highest phase achieved by the child and moves on to the next item card, through all 13 items. Items are then summed into a summary Peds NRS score using an algorithm.
Pediatric Evaluation of Disability Inventory (PEDI-CAT) | 6.5 months
  Pediatric Evaluation of Disability Inventory:
Pediatric Quality of Life Inventory CP Module (PedsQL-CP) | 6.5 months
  For each of the 4 domains, in addition to scaled scores, normative standard scores (provided as T-scores and age percentiles) are calculated. Normative scores describe the child's performance in comparison to other children of the same age (in one year intervals). For T-scores, the mean for each age group is 50, with a standard deviation of 10 (same format used for normative scores in the original PEDI). Typically, T-scores between 30 and 70 (i.e. mean ± 2 standard deviations) are considered within the expected range for age. Scores below 30 indicate decreased functional ability compared to what is typically expected for that age range. Scores above 70 indicate scores above what is typically expected for that age range. Higher scores indicate better outcome.
Functional near-infrared spectroscopy | 6.5 months
  Non-invasive, continuous wave functional near-infrared spectroscopy using an OctaMon+ (Artinis Medical Systems, Lieden, Netherlands) to identify metabolic changes and track oxygenation status.
Electromyography | 6.5 months
  Electrodes will measure voluntary (child is asked to perform a movement) and reflex activities (patellar reflex, achilles reflex, triceps reflex) of the dominant limbs.
ActiGraph sensors | 6.5 months
  Activity performance will be measured using ActiGraph accelerometers, which are motion sensors worn as a bracelet around the rist designed to detect movement when worn. They have excellent inter-instrument reliability (ICC = 0.98).

CONTACTS AND LOCATIONS:
Overall Officials: Megan B Flores, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No